CLINICAL TRIAL: NCT05391204
Title: Reproducibility of Strength Testing and Functional Testing of the Hip for the Return to Sport of Patients Activated by a Femoroacetabular Impingement: Comparison Between a Group of Patients and a Group of Healthy Controls
Acronym: H-Repro
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Ramsay santé (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-A01382-37
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-03

CONDITIONS: Femoroacetabular Impingement
Keywords: femoroacetabular Impingement; Reproducibility of strength testing and functional testing
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Intervention Model Description: There is therefore a lack of specific clinical tests allowing the functional evaluation of the hip. This is why it is necessary to study the possibility of deploying tests evaluating the functional capacities of the lower limb to characterize the functions of the hip.
  The study will compare patients group versus healthy volunteers and reproducibility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (Active Comparator): To answer the question of reproducibility of the measurement (1st objective), half of the group control will carry out two handover of the battery of functional tests to a week apart.
  Interventions: Other: Functional Tests
- Patients Volunteers (Experimental): To answer the question of reproducibility of the measurement (1st objective), half the group patient will perform two examinations at two months apart.
  Interventions: Other: Functional Tests

INTERVENTIONS:
Other: Functional Tests — Various physical exercices of inferior members

SUMMARY:
Reproducibility of strength testing and functional testing of the hip for the return to sport of patients activated by a femoroacetabular impingement: comparison between a group of patients and a group of healthy controls Femoroacetabular impingement is a disorder movement-related hip clinic, with bone abnormality at the joint coxo-femoral associated with a triad of symptoms, clinical signs and findings imagery. It represents premature contact symptomatic between the femur and the acetabulum. Currently, there is no consensus for determine when to return to sport securely after processing arthroscopy of a emoroacetabular impingement. Various clinical tests are used to assess the mobility or pain but no test studies specifically the level of recovery functional.

DETAILED DESCRIPTION:
Reproducibility of strength testing and functional testing of the hip for the return to sport of patients activated by a femoroacetabular impingement: comparison between a group of patients and a group of healthy controls Femoroacetabular impingement is a disorder movement-related hip clinic, with bone abnormality at the joint coxo-femoral associated with a triad of symptoms, clinical signs and findings imagery. It represents premature contact symptomatic between the femur and the acetabulum. Currently, there is no consensus for determine when to return to sport securely after processing arthroscopy of a emoroacetabular impingement. Various clinical tests are used to assess the mobility or pain but no test studies specifically the level of recovery functional.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Male or female aged 16 to 50
* Occurrence of the injury requiring surgery during a sports activity
* Hip arthroscopy
* Surgery performed by surgeons from the Santy Orthopedic Center (Lyon)
* Angle Alpha > 55°
* Patient having signed an informed consent
* Affiliated subject or beneficiary of a social Security

Control group

* Male or female aged 16 to 50
* Practicing a regular sporting activity In both groups
* Patient having signed an informed consent
* Affiliated subject or beneficiary of a social Security

Exclusion Criteria:

Patient group

* Contraindication of the surgeon
* Present another pathology of the hip on the side of the operated limb or on the contralateral side

Control group

* Declare a history of lower limb pain/injury in the last 12 months
* Declare a history of orthopedic surgery on the lower limbs

In any case will be excluded Protected subject: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Reproducibility rate | 8 months
  intra- and inter-session reproducibility

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu THAUNAT, Dr, Principal Investigator — Centre santy
Locations (1):
- Centre Santy, Lyon, AURA, France

IPD SHARING:
Plan to Share IPD: Undecided